CLINICAL TRIAL: NCT04126538
Title: Pirfenidone Capsule in Patients With Chronic Kidney Disease G2 and G3a Study on Safety and Pharmacokinetics of Single Dose
Brief Title: Pirfenidone Capsule in Patients With Chronic Kidney Disease G2 and G3a Study on Safety and Pharmacokinetics
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GNI-F647-1703
Record Dates: First submitted 2019-10-10; First posted 2019-10-15 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2021-03

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — pirfenidone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient group (Experimental): Patients with chronic kidney disease take pirfenidone capsule 400mg once orally
  Interventions: Drug: pirfenidone capsule
- Control group (Experimental): Healthy subjects take pirfenidone capsule 400mg once orally
  Interventions: Drug: pirfenidone capsule

INTERVENTIONS:
Drug: pirfenidone capsule — In the patient group, pirfenidone capsule was taken orally once for 400mg
  Arms: Patient group
Drug: pirfenidone capsule — Healthy subjects took pirfenidone capsule 400mg once orally
  Arms: Control group

SUMMARY:
To evaluate the safety and pharmacokinetic characteristics of pirfenidone capsules in chronic kidney disease G2 and G3a patients, and to provide a basis for the phase II clinical trial program

ELIGIBILITY:
Inclusion Criteria:

1. patients with chronic kidney disease, both male and female（Patient group）;
2. 18-70 years old, including 18 years old and 70 years old（Patient group）;
3. weight: male ≥50kg, female ≥45kg, 18≤BMI≤26 (BMI= weight (kg)/height 2 (m2))（Patient group）;
4. the stage of chronic kidney disease was G2 or G3a, indicating mild or moderate decrease in GFR, i.e., glomerular filtration rate was 45≤eGFR(ml/min/1.73m2) ≤89 (calculated according to ckd-epi formula)（Patient group）;
5. from 24h before the start of the study to the end of the study, subjects who agree to abstain from tobacco, alcohol, fruit juice, caffeine and tea（Patient group）;
6. I have had a detailed understanding of the nature, significance, possible benefits, possible inconvenience and potential risks of the trial before the study, and I have volunteered to participate in the clinical trial. I am able to communicate well with the investigator, comply with the requirements of the whole study, and have the ability to understand and sign the written informed consent.（Patient group）;
7. gender: Chinese healthy subjects, male and female（Control group）;
8. 18-70 years old, including 18 years old and 70 years old（Control group）;
9. weight: male ≥50kg, female ≥45kg, 18≤BMI≤26 (BMI= weight (kg)/height 2 (m2))（Control group）;
10. from 24h before the start of the study to the end of the study, subjects who agree to abstain from tobacco, alcohol, fruit juice, caffeine and tea（Control group）;
11. those who have detailed understanding of the nature, significance, potential benefits, possible inconveniences and potential risks of the trial before the study, who have volunteered to participate in the clinical trial, who can communicate well with the investigator, comply with the requirements of the whole study, and who are able to understand and sign a written informed consent（Control group）;

Exclusion Criteria:

1. （Physician visits） have participated in any other clinical trials within the first three months of the trial（Patient group）;
2. (preliminary) of any process may affect test security, or drug in the body of the disease, not including chronic kidney disease (CKD), including but not limited to: heart, liver, gastrointestinal tract, immune system and respiratory system always or the existing system diseases (especially for any impact on drug absorption of gastrointestinal diseases (such as irritable bowel syndrome symptoms, bowel disease or inflammatory bowel disease), active pathological bleeding (such as peptic ulcer), urticaria, eczema, dermatitis, epilepsy, allergic rhinitis, asthma, etc.)（Patient group）;
3. (consultation) allergy: if there are two or more drugs, food allergy history (including experimental drugs), lactose intolerance（Patient group）;
4. (consultation) any drugs that inhibit or induce drug metabolism in the liver (common liver enzyme inducers: barbiturates, carbamazepine, aminoximate, griseofulvin, aminopropyl, phenytoin, gromitol, rifampin, dexamethasone; Common liver enzyme inhibitors: chlorpromazine, cimetidine, ciprofloxacin, metronidazole, chloramphenicol, isoniazid, sulfonamide)（Patient group）;
5. (consultation) failure to follow a uniform diet (such as intolerance to standard meals, etc.) or difficulty swallowing（Patient group）;
6. (consultation) unable to tolerate venipuncture and/or having a history of blood or acupuncture（Patient group）;
7. (consultation) patients who have been drinking excessive amounts of tea, coffee or caffeinated drinks (more than 8 cups a day, 1 cup =250mL) for a long time; Or taking any food or beverage containing caffeine (such as coffee, strong tea, chocolate, etc.) within 24 hours before the first administration of the drug（Patient group）;
8. (consultation) previous binge drinking (i.e., male drinking more than 28 units per week and female drinking more than 21 units per week (1 unit contains 14g alcohol, such as 360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine); Or who had regularly consumed alcohol (more than 14 units per week) during the 6 months prior to the trial; Or who had taken any alcoholic product within 24 hours of initial administration（Patient group）;
9. (consultation) those who had donated blood or suffered massive bleeding (greater than 450 mL) within 3 months before the first administration of the study, or who planned to donate blood or blood components during the study period or within 3 months after the end of the study（Patient group）;
10. (consultation) acute disease during the screening phase before study or before study medication（Patient group）;
11. (consultation) patients who had taken food or drinks containing enzymes that can induce or inhibit liver metabolism (e.g., grapefruit, mango, pitaya, grape juice, orange juice, etc., rich in flavonoids or citrus glycosides) within 24 hours before the first administration were studied（Patient group）;
12. pregnant or lactating women, and subjects (or their partners) who have a pregnancy plan during the trial and within 3 months after the end of the study and who do not agree to use non-drug contraception during the trial（Patient group）;
13. (consultation) those who have had surgery within three months before the screening period, or who are planning to have surgery during the study period, and those who have had surgery that will affect drug absorption, distribution, metabolism and excretion（Patient group）;
14. (consultation) previous history of drug abuse or drug abuse（Patient group）;
15. (consultation) persons who have smoked more than 5 cigarettes per day in the 14 days before screening, or who cannot stop using any tobacco products during the trial（Patient group）;
16. screening for smoking or using any tobacco products up to admission（Patient group）;
17. screening phase physical examination, vital signs measurement, electrocardiogram examination, laboratory examination (hematuria routine, blood coagulation function, blood pregnancy (women of childbearing age only)) and investigator determination of clinically significant abnormalities (excluding abnormalities caused by chronic kidney disease). Abnormal liver function examination (ALT, AST, ALP, gamma GT, TP, Alb, A/G, t-bil, d-bil) suggested liver disease or liver injury. Renal function test SCr > 400 mol/L; Abnormal blood electrolyte examination (K+, Na+, Cl-, Ca2+) suggested high potassium or acidosis.（Patient group）
18. nicotine positive test（Patient group）;
19. alcohol breath test with test results greater than 0.0mg/100ml（Patient group）;
20. positive urine drug screening（Patient group）;
21. hepatitis b surface antigen positive, or hepatitis c antibody positive, or syphilis spirochete antibody positive, or HIV antibody positive（Patient group）;
22. the investigator considers that there are any circumstances that may affect the subject's informed consent or adherence to the study protocol, or participation in the study may affect the study results or their own safety.（Patient group）;
23. （Physician visits）those who participated in any other clinical trials three months prior to the trial（Control group）;
24. (preliminary) of any process may affect test security, or drug in the body of the disease, including but not limited to: heart, liver, kidney, endocrine, the digestive tract, immune system and respiratory system always or the existing system diseases (especially cardiovascular diseases including cardiovascular disease risk, any impact on drug absorption of gastrointestinal diseases (such as irritable bowel syndrome symptoms, bowel disease or inflammatory bowel disease), active pathological bleeding (such as peptic ulcer), urticaria, eczema, dermatitis, epilepsy, allergic rhinitis, asthma, etc.)（Control group）;
25. (consultation) allergy: if there are two or more drugs, food allergy history (including experimental drugs), lactose intolerance（Control group）;
26. (consultation) any drugs that inhibit or induce drug metabolism in the liver (common liver enzyme inducers: barbiturates, carbamazepine, aminoximate, griseofulvin, aminopropyl, phenytoin, gromitol, rifampin, dexamethasone; Common liver enzyme inhibitors: chlorpromazine, cimetidine, ciprofloxacin, metronidazole, chloramphenicol, isoniazid, sulfonamide); Or have used any medicines (including Chinese herbal medicines) or health supplements within 14 days prior to initial administration（Control group）;
27. (consultation) failure to follow a uniform diet (such as intolerance to standard meals, etc.) or difficulty swallowing（Control group）;
28. (consultation) unable to tolerate venipuncture and/or having a history of blood or acupuncture（Control group）;
29. (consultation) patients who have been drinking excessive amounts of tea, coffee or caffeinated drinks (more than 8 cups a day, 1 cup =250mL) for a long time; Or taking any food or beverage containing caffeine (such as coffee, strong tea, chocolate, etc.) within 24 hours before the first administration of the drug（Control group）;
30. (consultation) previous binge drinking (i.e., male drinking more than 28 units per week and female drinking more than 21 units per week (1 unit contains 14g alcohol, such as 360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine); Or who had regularly consumed alcohol (more than 14 units per week) during the 6 months prior to the trial; Or who had taken any alcoholic product within 24 hours of initial administration（Control group）;
31. (consultation) those who had donated blood or suffered massive bleeding (greater than 450 mL) within 3 months before the first administration of the study, or who planned to donate blood or blood components during the study period or within 3 months after the end of the study（Control group）;
32. (consultation) acute disease during the screening phase before study or before study medication（Control group）;
33. (consultation) patients who had taken food or drinks containing enzymes that can induce or inhibit liver metabolism (e.g., grapefruit, mango, pitaya, grape juice, orange juice, etc., rich in flavonoids or citrus glycosides) within 24 hours before the first administration were studied（Control group）;
34. pregnant or lactating women, and subjects (or their partners) who have a pregnancy plan during the trial and within 3 months after the end of the study and who do not agree to use non-drug contraception during the trial（Control group）;
35. (consultation) those who have had surgery within three months before the screening period, or who are planning to have surgery during the study period, and those who have had surgery that will affect drug absorption, distribution, metabolism and excretion（Control group）;
36. (consultation) previous history of drug abuse or drug abuse（Control group）;
37. (consultation) persons who have smoked more than 5 cigarettes per day in the 14 days before screening, or who cannot stop using any tobacco products during the trial（Control group）;
38. screening for smoking or using any tobacco products up to admission（Control group）;
39. screening phase physical examination, vital signs measurement, electrocardiogram examination, b-mode ultrasound examination, laboratory examination [blood routine, urine routine, blood biochemistry, blood coagulation function, blood pregnancy (women of childbearing age only)], and the investigator judged that abnormalities were clinically significant（Control group）;
40. those with positive nicotine test results（Control group）;
41. alcohol breath test with test results greater than 0.0mg/100ml（Control group）;
42. positive urine drug screening（Control group）;
43. hepatitis b surface antigen positive, or hepatitis c antibody positive, or syphilis spirochete antibody positive, or HIV antibody positive（Control group）;
44. the investigator considers that there are any circumstances that may affect the subject's informed consent or adherence to the study protocol, or participation in the study may affect the study results or their own safety.（Control group）.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-08-27 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Plasma drug concentrations of pirfenidone | up to 24 weeks
Urine concentration of pirfenidone | up to 24 weeks

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shaojun Shaojun, Doctor, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China